CLINICAL TRIAL: NCT03225781
Title: A Clinical Trial Using Electrochemotherapy With Bleomycin for the Treatment of Non-metastatic Unresectable Pancreatic Cancer
Brief Title: Electrochemoterapy With Bleomycin for the Treatment of Unresectable Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic reasons
Sponsor: Universita di Verona (Other)
Collaborators: IGEA (Industry)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, MD, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-ECT
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrochemotherapy with Bleomycin — Application of Reversible Electroporation (Electrochemotherapy) with Bleomycin

SUMMARY:
Electrochemotherapy is a type of electroporation that allows the delivery of drugs to the cells through the local creation of pores in the cell membrane. The electric pulses can be applied directly to the neoplastic cells, allowing for the local concentration of a possible chemotherapeutic agent administered through the bloodstream. This technique does not use heat nor other thermal energies and it is performed using special needles/electrodes linked to a generator ("porator").

In this study this technique will be applied on unresectable pancreatic cancer, already submitted to neoadjuvant treatment and still unresectable, through laparotomy. Bleomycin will be the chemotherapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

* Radiologic confirmation of locally advanced pancreatic cancer by at least contrast enhanced CT of chest and abdomen (with the upper abdomen scanned according to a dedicated 3mm slice multiphase pancreatic tumor protocol), performed maximum 4 weeks prior to the procedure
* Cytohistological diagnosis of pancreatic cancer
* Age > 18 and < 80
* Stable disease after chemotherapy (no tumor progression, no oncomarkers (Carbohydrate Antigen 19-9 [CA 19-9] or Carcinoembryonic antigen [CEA]) increase
* Performance Status 0 sec. ECOG (Eastern Cooperative Oncology Group)
* Written informed consent

Exclusion Criteria:

* Resectable pancreatic cancer as assessed by multidisciplinary meeting
* Stage IV disease
* Patients receiving fenitoin, phosphofenitoin or living vaccines
* Pregnancy
* Progressive disease (either dimensional and not only by stage)
* < 18 years old and > 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, 1 year
  Number of adverse events related with electrochemotherapy (within 12 months after treatment) are registered and analyzed according to the CTCAE version 4.0. Complications are distinct in early (during hospitalization) and late (bile duct stenosis) that may appear during follow-up

SECONDARY OUTCOMES:
Feasibility | through study completion, 1 year
  Number of procedures planned actually performed
Tumour response | 12 months
  Analysis of effects of electrochemotherapy on tumor using RECIST criteria
Quality of life | 12 months
  Analysis of quality of life using the Karnovsky performance index
Quality of life | 12 months
  Analysis of quality of life using the pain numeric scale
Survival | 12 months
  Survival analysis through the calculation of overall survival
Survival | 12 months
  Survival analysis through the calculation of progression free survival survival
Immunomonitoring | From baseline to the first month
  Study of adaptive immunity through the sampling of Interleukin6 and Heat shock protein 70 levels at baseline and post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona Hospital, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Granata V, Fusco R, Piccirillo M, Palaia R, Petrillo A, Lastoria S, Izzo F. Electrochemotherapy in locally advanced pancreatic cancer: Preliminary results. Int J Surg. 2015 Jun;18:230-6. doi: 10.1016/j.ijsu.2015.04.055. Epub 2015 Apr 24. PMID 25917204
- [Result] Bimonte S, Leongito M, Granata V, Barbieri A, Del Vecchio V, Falco M, Nasto A, Albino V, Piccirillo M, Palaia R, Amore A, Giacomo Rd, Lastoria S, Setola SV, Fusco R, Petrillo A, Izzo F. Electrochemotherapy in pancreatic adenocarcinoma treatment: pre-clinical and clinical studies. Radiol Oncol. 2016 Feb 16;50(1):14-20. doi: 10.1515/raon-2016-0003. eCollection 2016 Mar 1. PMID 27069445
- [Result] Campana LG, Mocellin S, Basso M, Puccetti O, De Salvo GL, Chiarion-Sileni V, Vecchiato A, Corti L, Rossi CR, Nitti D. Bleomycin-based electrochemotherapy: clinical outcome from a single institution's experience with 52 patients. Ann Surg Oncol. 2009 Jan;16(1):191-9. doi: 10.1245/s10434-008-0204-8. Epub 2008 Nov 6. PMID 18987914
- [Result] Girelli R, Prejano S, Cataldo I, Corbo V, Martini L, Scarpa A, Claudio B. Feasibility and safety of electrochemotherapy (ECT) in the pancreas: a pre-clinical investigation. Radiol Oncol. 2015 Mar 25;49(2):147-54. doi: 10.1515/raon-2015-0013. eCollection 2015 Jun. PMID 26029026